CLINICAL TRIAL: NCT01221155
Title: Extending Ultrasound Elastography to Manual Treatment Methods
Status: Completed | Type: Observational
Sponsor: Canadian Memorial Chiropractic College (Other)
Responsible Party: Sponsor
Other Study IDs: 72152
Record Dates: First submitted 2010-09-23; First posted 2010-10-14 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Back Pain
Keywords: Musculoskeletal
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Manual treatment offers benefit to some patients suffering from back pain but little is known about which of the many tissue layers are affected. This study will help identify which tissues may be stimulated sufficiently to be a source for the clinical effects of treatment and to prioritize future work to understand mechanisms of back pain and to improve care.

Current soft-tissue ultrasound elastography techniques, under static condition, will be extended to quantify relative displacement and strains(active and passive)across the depth of tissue strata that arise from small amplitude motions during continuous passive motion clinical procedures and in weight bearing postures. Relative movement of the stratified layers of the back, from treatment and task-generated perturbations, will enable the elastography interrogation of the tissue.

DETAILED DESCRIPTION:
1. Tissue displacement and strain differs dependent on comparable tasks, in recumbent vs upright postures and muscular activation.

   - Refine motion tracking and stabilization of manual elastography, used in preliminary study, to evaluate layered tissue strain patterns during clinical continuous passive motion (flexion, extension and lateral bending) and standardized weight bearing (stance, flexion to 15 degrees and arm-extended weight holding).
2. Relative muscle activity is significantly related to muscle strain ratio.

   - Evaluate the biceps as a simple model, in parallel, for displacement and elastography changes.
3. Displacement and strain decrease monotonically as depth of paraspinal tissue from the surface increases.

   - Evaluate the timing relationship of total passive loads, myoelectric paraspinal behavior displacement/strain characteristics at the l4/l5 level for the longissimus, intermuscular fascia and multifidus at baseline and during standardize weight bearing tasks as well as at recumbent baseline, during and return to neutral for prone and lateral recumbent continuous passive motion maneuvers.
4. Change in tissue displacement and strains differ between healthy and unhealthy individuals when change in muscle activity and tissue layer are taken into account.

   * Assess any differences in displacement and strain characteristics of the layered longissimus, intermuscular fascia and multifidus between healthy and chronic low back patients in the timing relationship to movement, total passive load amplitudes and myoelectric activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* a clean history
* no episode of disabling back pain
* no episode of disabling leg pain
* no episode within the prior 90 days will be required Back Pain Subjects
* experiencing continuous episodes of low back pain within the prior 90 days
* experiencing recurring episodes of low back pain within the prior 90 days
* have pain at >3.0 on Visual Analogue Scale

Exclusion Criteria:

* history of diabetes
* history of neuromuscular disease
* history of scoliosis apparent on inspection
* a bleeding disorder
* collagen vascular disease
* corticosteroid therapy
* extensive scarring or dermatological abnormalities, including adhesive tape sensitivity
* women who are pregnant or have active menstruation will be excluded to avoid positional discomfort.
* pain radiating below the knee or loss of motor, bowel or bladder control

Volunteers taking anti-inflammatory or antihistamine medications will be asked to discontinue their use 3 days before testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1: Fifteen healthy volunteers from Canadian Memorial Chiropractic College (CMCC) community.
  Group 2: 30 Subjects (15 healthy volunteers and 15 chronic low back pain)
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2007-12; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The quantitative tissue displacement and strains. | baseline and 6 weeks
  These parameters may be considered as total cumulative displacement and strain over the recording interval or smaller epochs sequentially over time. After analysis completion, power and effect sizes will be calculated for the various parameters being studied. In cases where statistical power is found to be insufficient, calculation for appropriate sample size estimates will be compiled to guide future work. Secondary analyses will explore linear vs non-linear representations of the data. The best fit of linear/nonlinear correlations will be used to describe all muscle relationships.
Timing of change in the relative myoelectric activity. | baseline and 6 weeks
  These parameters may be considered as total cumulative displacement and strain over the recording interval or smaller epochs sequentially over time. After analysis completion, power and effect sizes will be calculated for the various parameters being studied. In cases where statistical power is found to be insufficient, calculation for appropriate sample size estimates will be compiled to guide future work. Secondary analyses will explore linear vs non-linear representations of the data. The best fit of linear/nonlinear correlations will be used to describe all muscle relationships.
Strain ratio in the context of a series of motions in upright/recumbent postures and in healthy/chronic low back pain volunteers. | baseline and 6 weeks
  These parameters may be considered as total cumulative displacement and strain over the recording interval or smaller epochs sequentially over time. After analysis completion, power and effect sizes will be calculated for the various parameters being studied. In cases where statistical power is found to be insufficient, calculation for appropriate sample size estimates will be compiled to guide future work. Secondary analyses will explore linear vs non-linear representations of the data. The best fit of linear/nonlinear correlations will be used to describe all muscle relationships.

CONTACTS AND LOCATIONS:
Overall Officials: John J. Triano, DC, PhD, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada